CLINICAL TRIAL: NCT00753805
Title: Dietetic Effects of Oral Intervention With Mare's Milk on the SCORAD, Faecal Microbiota and Immunological Parameters in Patients With Atopic Dermatitis
Brief Title: Dietetic Effects of Mare's Milk in Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. G. Jahreis, University of Jena, Dept. of Nutritional Physiology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSEP H15-04
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-06

CONDITIONS: Atopic Dermatitis
Keywords: mare's milk; atopic dermatitis; endogenous eczema; SCORAD; Bifidobacteria
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: mare's milk — The participants received 250 ml mare's milk or placebo daily. The placebo drink was based on a hypoallergenic infant formula.

SUMMARY:
The study was performed to investigate the effects of mare's milk on SCORAD, faecal microbiota and immunological parameters in patients with atopic dermatitis.

DETAILED DESCRIPTION:
Mare's milk has been used in the treatment of inflammatory illnesses for centuries since it was known to contain antimicrobial, anti-inflammatory and immunomodulatory substances. The aim of this study was to examine whether the consumption of mare's milk by patients with atopic dermatitis (AD) has a beneficial effect.

As a precondition for participating in this study, the subjects were provided information in writing and verbally about the details of the study. Informed consent was obtained from all volunteers. Before the beginning of the study, all participants were subject to a medical examination in the Clinic for Dermatology and Dermatologic Allergology of the Friedrich Schiller University Jena. The AD was diagnosed according to the atopy-score of Diepgen. Severity of eczema was evaluated by using the SCORAD score. A skin prick test was performed for the exclusion of type 1 sensitivity to mare's milk.

The study was designed as a double blind, placebo-controlled crossover trial. Twenty-three patients received 250-ml mare's milk or placebo orally for 16 consecutive weeks. Between the two intervention periods, a four week wash-out period without drinking any test substances was introduced. The intensity of AD was examined using the Severity Scoring of Atopic Dermatitis (SCORAD), which was determined at the start of the study and after 4, 8, 12 and 16 weeks of each intervention period. Blood samples were taken at the start of the study and subsequently after 8 and 16 weeks. Fresh stool samples were taken at the beginning of the study and at the end of each intervention period.

ELIGIBILITY:
Inclusion Criteria:

* A clear and definite diagnosis of AD
* Willingness to use only the recommended drugs
* Competence regarding the daily documentation of skin state and well being.

Exclusion Criteria:

* Therapy with non recommended drugs one month before start of the study
* Active skin infection
* Apparent asthma
* Intolerance against milk
* Long-term therapy with drugs
* Symptomatic heart disease and/or internal disease
* Autoimmune diseases, immune defects, and malignoma
* Alcohol and drug abuse.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2004-08; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
SCORAD change | 16 weeks

SECONDARY OUTCOMES:
Immunological parameters (ECP, sE-selectin, MDC, IL-16), inflammation biomarker CRP, selected faecal microbiota (bifidobacteria, lactobacilli) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — University of Jena, Dept. of Nutritional Physiology
Locations (1):
- University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia, Germany